CLINICAL TRIAL: NCT03314129
Title: Visual Remediation in Schizophrenia
Brief Title: Remediation of Visual Perceptual Impairments in People With Schizophrenia
Acronym: VRiS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: New York University (Other); Weill Medical College of Cornell University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Steven Silverstein, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20170000922; R61MH115119 (NIH)
Record Dates: First submitted 2017-10-04; First posted 2017-10-19 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Contrast sensitivity (Experimental): UltimEyes
  Interventions: Behavioral: UltimEyes
- Perceptual organization (Experimental): Contour Integration Training
  Interventions: Behavioral: Contour Integration Training
- Contrast sensitivity + Perceptual org. (Experimental): UltimEyes + Contour Integration Training
  Interventions: Behavioral: UltimEyes + Contour Integration Training
- Cognitive remediation (Active Comparator): MyBrainSolutions
  Interventions: Behavioral: MyBrainSolutions

INTERVENTIONS:
Behavioral: UltimEyes — A computer program developed to improve contrast sensitivity and visual acuity.
  Arms: Contrast sensitivity
Behavioral: Contour Integration Training — A computerized program to improve contour integration (a form of perceptual organization).
  Arms: Perceptual organization
Behavioral: UltimEyes + Contour Integration Training — The combination of UltimEyes and Contour Integration Training
  Arms: Contrast sensitivity + Perceptual org.
Behavioral: MyBrainSolutions — A computer program consisting of exercises to improve cognition (attention, memory, planning) and to facilitate goal setting.
  Arms: Cognitive remediation

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a visual remediation intervention for people with schizophrenia. The intervention targets two visual functions that much research has shown are impaired in many people with the disorder, namely contrast sensitivity and perceptual organization. The first phase of the study will test the effects of interventions targeting each of these processes, as well as the effects of a combined package. A control condition of higher-level cognitive remediation is included as a fourth condition. The second phase of the study will evaluate the effectiveness of the most effective intervention from the first phase, but in a new and larger sample of individuals. Outcome measures include multiple aspects of visual functioning, as well as visual cognition and overall community functioning.

DETAILED DESCRIPTION:
It is increasingly clear that people with schizophrenia have a range of visual perception impairments, including in low-level vision (e.g., acuity, contrast sensitivity) and mid-level vision (e.g., perceptual organization, coherent motion detection). These impairments are significantly related to poorer performance on cognitive (e.g., visual learning and memory) and social cognitive (e.g., facial emotion decoding) measures, and to worse functional outcomes. To date, there is no accepted technique for visual remediation for schizophrenia, and almost no work has been done in this area. However, visual remediation is a well-developed subfield within cognitive rehabilitation for traumatic brain injury (TBI) patients, and initial studies of short-term visual perceptual learning in schizophrenia indicate that plasticity exists that could support longer-term changes. Therefore, the overall goal of the proposed project is to test a visual remediation intervention for schizophrenia and determine its effects on specific visual targets with well-understood neurobiological mechanisms. The goal of the R61 is to determine the optimal intervention for improving the targets of contrast sensitivity (CS) and perceptual organization (PO). Extensive evidence exists for impaired CS and PO in schizophrenia. Moreover, these targets are prototypical examples of gain control and integration, respectively, which were identified by the NIMH-sponsored CNTRICS initiative as being the two core mechanisms involved in visual disturbances in the disorder. The investigators will examine two computer-based interventions. One, ULTIMEYES (UE), targets CS. The other, contour integration training (CIT), targets PO. The investigators will also examine the effects of combined treatment (UE&CIT). An active computer-based control treatment will be included. There will be 40 sessions, with assessments after every 10 sessions (N=20/group). The R61 Specific Aim is to evaluate the effects of UE and CIT on CS and PO targets, respectively, to determine if treatment effects meet a pre-specified effect-size criterion. Results of the R61 will be used to identify the treatment (UE, CIT, or UE&CIT) and duration (i.e., dose) that most effectively and efficiently improves the target(s). The goal of the R33 is to conduct an initial randomized controlled trial (RCT) of the optimal treatment identified in the R61. The R33 Specific Aims are to: 1) replicate and extend R61 results supporting visual target engagement in an adequately powered RCT (N=50/group); and 2) determine if visual target engagement is associated with improvements in cognition, social cognition, and functional capacity. If the R33 hypotheses are confirmed, results will inform the design of a later RCT to further explore mediators and moderators of treatment effects, and to move towards a precision medicine approach, wherein we determine which individuals are most likely to benefit from this intervention.

ELIGIBILITY:
Inclusion Criteria:

1. SCID-5 diagnosis of schizophrenia;
2. 18-60 years old;
3. speaks English;
4. able to complete the MATRICS Consensus Cognitive Battery (MCCB) at the baseline assessment (for R33);
5. a raw score of 37 or greater on the Wide Range Achievement Test, Reading subtest (WRAT-3), to establish a minimum reading level (6th grade) and to estimate premorbid IQ; and
6. clinically stable as indicated by no antipsychotic medication changes in the last month or if on depot, no change in the past 2 months.

Exclusion Criteria:

1. history of intellectual disability, or developmental or neurological disorder;
2. history of brain trauma associated with loss of consciousness for > 10 minutes or behavioral sequelae;
3. alcohol or substance use disorder within the last 6 months; and
4. history of eye disease (e.g., glaucoma, retinopathy).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Contrast sensitivity - behavioral | Years 1-5
  Peak contrast, as measures by a behavioral (psychophysical) measure of contrast sensitivity.
Contrast sensitivity - electrophysiological | Years 1-5
  Steady state visual evoked potential (ssVEP) amplitudes recorded during the contrast sensitivity task.
Contour integration | Years 1-5
  Total score on the Jittered-Orientation Visual Integration Task, or JOVI), a psychophysical measure of perceptual organization.

SECONDARY OUTCOMES:
Reading speed | Years 3-5
  Minnesota Low-Vision Reading Test (MNREAD): This test assesses reading speed ability. The charts contain 19 English sentences (60 characters each) with print sizes ranging from 1.3 to -0.5 logMAR at a distance of 16 inches (0.41 meters).
Emotion recognition | Years 3-5
  Total score on the Penn Emotion Recognition Test, a computerized test of emotion recognition.
Cognition | Years 3-5
  Total score on the MATRICS Consensus Cognitive Battery
Community functioning | Years 3-5
  Total score on the UCSD Performance-Based Skills Assessment (UPSA), a test of the ability to perform various skills important in residential and community settings.

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Silverstein, Ph.D., Principal Investigator — University of Rochester
Locations (2):
- United States (2):
  - University of Rochester Medical Center - Strong Ties Community Support Clinic, Rochester, New York
  - New York Presbyterian Hospital, White Plains, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silverstein SM, Seitz AR, Ahmed AO, Thompson JL, Zemon V, Gara M, Butler PD. Development and Evaluation of a Visual Remediation Intervention for People with Schizophrenia. J Psychiatr Brain Sci. 2020;5:e200017. doi: 10.20900/jpbs.20200017. Epub 2020 Jul 20. PMID 32789191
- [Result] Butler PD, Thompson JL, Seitz AR, Deveau J, Silverstein SM. Visual perceptual remediation for individuals with schizophrenia: Rationale, method, and three case studies. Psychiatr Rehabil J. 2017 Mar;40(1):43-52. doi: 10.1037/prj0000212. Epub 2016 Aug 22. PMID 27547852

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-13): https://cdn.clinicaltrials.gov/large-docs/29/NCT03314129/Prot_SAP_000.pdf